CLINICAL TRIAL: NCT06277596
Title: Comparison of the Effects of Progressive Clinical Pilates Exercises Applied as a Supervised and Home Program in Individuals With Fibromyalgia
Brief Title: The Effects of Progressive Clinical Pilates Exercises Applied as 2 Different Ways in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-2023-0101
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia
Keywords: Exercise; chronic pain; clinical pilates; Functional; Psychosocial
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervise clinical Pilates group (Experimental): Clinical Pilates exercises will be performed 10 repetitions, 3 days a week, for 6 weeks, under the supervision of a physiotherapist. The exercise program will be progressed as basic stabilization exercises in the first 3 weeks, advanced stabilization exercises in the last 3 weeks, as recommended in the literature, and a 30-second rest will be given between sets.
  Interventions: Other: Exercise
- Clinical Pilates as home exercise (Active Comparator): The same exercises will be shown to the home exercise group and it will be ensured that they are performed correctly. Patients will be given an illustrated and descriptive exercise program brochure containing information about exercise position, number of repetitions, contraction duration, rest time between sets, frequency, and an exercise diary for exercise tracking. In the 3rd week, new exercises will be shown to individuals. It will be applied 10 times, 3 days a week, for 6 weeks. The exercise program will be progressed as basic stabilization exercises in the first 3 weeks, advanced stabilization exercises in the last 3 weeks, as recommended in the literature, and a 30-second rest will be given between sets.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Clinical Pilates exercises (basic and advanced stabilization exercises)

SUMMARY:
The aim of this study is to compare the effects of progressive clinical Pilates exercises applied as group under the supervision of a physiotherapist and home exercise programs on pain level, physical condition, functional status, psychosocial status and quality of life in individuals with fibromyalgia between the ages of 20-50.

DETAILED DESCRIPTION:
After the voluntary individuals with Fibromyalgia (FM) who meet the inclusion criteria are evaluated, they will be randomly divided into two groups: exercise group and home exercise group.

The same clinical Pilates program will be applied to both groups at the same dosage. Evaluations and treatment will be applied to both groups by the same physiotherapist. Individuals will perform the exercises 10 repetitions, 3 days a week, for 6 weeks. The exercise program will be progressed as basic stabilization exercises in the first 3 weeks, advanced stabilization exercises in the last 3 weeks, as recommended in the literature, and a 30-second rest will be given between sets. For the home exercise group, all exercises will be shown and it will be ensured that they are performed correctly. Patients will be given an illustrated and descriptive exercise program brochure containing information about exercise position, number of repetitions, contraction duration, rest time between sets, frequency, and an exercise diary for exercise tracking.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer individuals between the ages of 20-50
* Diagnosed with fibromyalgia according to the American College of Rheumatology criteria
* Pain level 3 and above according to visual analogue scale.
* Individuals who are sedentary (who have not engaged in physical activity at least 3 days a week in the last 3 months) will be included in the study.

Exclusion Criteria:

* Having additional rheumatic disease
* Using NSAIDs and antidepressant drugs
* Individuals with orthopedic, neurological and cardiopulmonary diseases that prevent them from exercising
* Pregnant women
* Malignancy
* Individuals with uncontrolled systemic diseases (diabetes, systemic arterial hypertension, thyroid dysfunction, neurological, cardiorespiratory, musculoskeletal problems, etc.)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale ( VAS ) | 6 weeks
  Pain during activities of daily living and at rest will be evaluated with the Visual Analogue Scale (VAS). The individual will be asked to mark the appropriate point on a 10-centimeter (cm) horizontal line between 0 (no pain) and 10 (unbearable pain) at both ends. The distance between the point marked by the individual and the start will be measured with a ruler in cm and recorded. A 2-point reduction in VAS is considered a clinically important improvement.

SECONDARY OUTCOMES:
Sociodemographic information (age) | 6 weeks
  Age will be recorded as years
Sociodemographic information (height) | 6 weeks
  Height will be measured and recorded as centimeters (cm)
Sociodemographic information (weight) | 6 weeks
  Weight will be measured and recorded as kilogram (kg)
Trunk Muscle Endurance (McGill Endurance Test and Plank Test) | 6 weeks
  McGill Endurance Test:
  * Lateral Bridge Test: used to evaluate trunk lateral muscle endurance. The time will be measured and recorded with a stopwatch in seconds. The test will be repeated once for the right and left sides.
  * Biering-Sorenson Test: It will be used to evaluate the static endurance of the back extensors.
  * Trunk flexor test: It will be used to evaluate the muscle endurance of the trunk flexors.
  Plank Test: It will be used to evaluate whole body muscle endurance. It has a high reliability of 95 %.
  For each test, the time until the body position is disrupted will be measured with a stopwatch and recorded in seconds.
Chair Sit to stand test | 6 weeks
  It will be used to evaluate lower extremity proximal muscle strength and endurance. The individual will sit in the middle of the chair with his back upright, his feet on the floor, and his arms crossed in front of his chest. By starting the time with a stopwatch, the individual will be asked to perform the full standing and sitting movement as many times as possible in 30 seconds and the number of full stands will be recorded.
6 minute walk test | 6 weeks
  It will be used to assess the functional capacity. At the end of the 6 minute, the distance walked will be recorded as meters (m).
Fatigue Severity Scale | 6 weeks
  It will be used to evaluate the effect of fatigue on functionality. In this scale, which evaluates individuals' fatigue level in the last week, the scores from the questions (1: strongly disagree, 7: strongly agree) will be summed and divided by the number of questions to calculate the total score. Scores of 4 and above indicate serious fatigue.
Pittsburgh Sleep Quality Index | 6 weeks
  Habitual sleep efficiency, sleep duration, use of sleeping pills, daytime dysfunction, sleep latency, sleep quality and sleep disturbance in the last month will be evaluated.
  The total score obtained from the index, which is scored between 0-3, varies between 0-21. A total score between 0 and 4 points indicates good sleep quality, while a total score between 5 and 21 points indicates poor sleep quality.
Revised Fibromyalgia Impact Questionnaire | 6 weeks
  Limitations and functional disability in individuals will be evaluated with this survey. The questionnaire consists of 21 questions and each question is evaluated on a numerical scale between 0-10. An increase in the score obtained from the survey indicates that the loss of function due to fibromyalgia (FM) increases.
Fear-Avoidance Beliefs Questionnaire | 6 weeks
  It consists of 2 parts including questions about physical activities and work. In the questionnaire evaluated with a 7-point Likert-type scale, physical activities are scored between 0-24, while work-related questions are scored between 0-36. A high score indicates that the individual has high fear avoidance beliefs.
Pain Self-Efficacy Questionnaire | 6 weeks
  It evaluates the degree of confidence in performing activities despite pain. It is a questionnaire that is practical due to its brevity (10 questions) and measures multiple domains of self-efficacy related to social and physical functions. It is a 7-point Likert-type scale. The total score ranges from 0 to 60, with higher scores indicating higher self-efficacy.
Body Awareness Questionnaire | 6 weeks
  Body image will be assessed with this questionnaire. It consists of 4 subgroups (prediction of body reactions, sleep-wake cycle, prediction at the beginning of the disease, and attention to changes and reactions in body processes). Participants will be asked to give points between 1 and 7 for each of the 18 statements. A high score means high body awareness.
Cognitive Exercise Therapy Approach-Biopsyhosocial Questionnaire (BETY-BQ) | 6 weeks
  This questionnaire which consists of 30 items, will be used to evaluate the biopsychosocial status of individuals. Each item is scored on a 5-point Likert-type scale that can be scored between 0 (no/never) and 4 (yes/always). The higher the total score, the higher the individual's biopsychosocial situation is.
Short form-36 (SF-36) | 6 weeks
  It will be used to assess the quality of life. It generally evaluates the perception of health, social and physical functions, vitality, mental health, role limitations due to physical and emotional distress, and body pain with a total of 36 items. Each title is calculated separately and scores are given between 0-100. A high score indicates good health and a low score indicates poor health.
Treatment Satisfaction Evaluation | 6 weeks
  To determine the treatment satisfaction level, the individual will be asked to mark between 0 (very dissatisfied) and 10 (extremely satisfied) on a 10 centimeter (cm) horizontal line. The distance between the marked location and point 0 was recorded in centimeter (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kadıoğlu, PT, Principal Investigator — Eastern Mediterranean University; Sevim Oksuz, Asst.Prof.Dr, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus